CLINICAL TRIAL: NCT02678611
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate Safety and Health Benefits of Basis™ Among Elderly Subjects.
Brief Title: A Study to Evaluate Safety and Health Benefits of Basis™ Among Elderly Subjects.
Acronym: 15BSHE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elysium Health (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 15BSHE
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Safety: Healthy Subjects
Keywords: Healthy participants; Dietary supplement; Safety; Tolerability; Older Adults; Basis; Nicotinamide riboside; Pterostilbene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Basis 250 (Experimental)
  Interventions: Dietary Supplement: Basis 250
- Basis 500 (Experimental)
  Interventions: Dietary Supplement: Basis 500
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Basis 250
  Arms: Basis 250
Dietary Supplement: Basis 500
  Arms: Basis 500
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the safety, tolerability and potential health benefits of the dietary supplement, Basis. There will be two doses of Basis compared to a placebo. One third of subjects will receive the low dose Basis, one third will receive the higher dose Basis and one third will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 60 to 80 (inclusive) years of age
* Body Mass Index (BMI) must be 18 to 35 kg/ m2 (±1 kg/m2)
* •Be able to make scheduled office visits 4 times during the study
* Willing to follow the instructions and complete multiple study questionnaires and assessments
* Agrees to avoid taking Vitamin B3 (Niacin, Nicotinic acid or niacinamide) supplements or multivitamins 14 days prior to randomization and for the duration of the study period
* Healthy otherwise as determined by laboratory results and medical history
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* History of any significant chronic disease or any clinically active illness within 3 months of study entry, including any history of renal or liver impairment, any endocrine, inflammatory, cardiovascular, gastro-intestinal, neurological, psychiatric, neoplastic or metabolic disease. Clinical significance of disease will be assessed by the Qualified Investigator and eligibility determined.
* Significant or untreated medical disorders including recent myocardial ischemia or infarction, unstable angina, uncontrolled hypertension, AIDS, malignancy, epilepsy, and recent cerebrovascular disease
* Subjects with or who have recently experienced a traumatic injury, infections or undergone surgery
* Subjects with history of pellagra or niacin deficiency
* Taking lipid lowering drugs
* Use of natural health products containing Nicotinamide riboside within 14 days prior to randomization and during the course of the study
* History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Volunteers with cancer in full remission more than 5 years after diagnosis are acceptable
* Has participated in any clinical trial with an investigational medicinal product within the past three months prior to the first dose in the current study
* Unstable medical conditions
* Alcohol use >2 standard alcoholic drinks per day
* History of alcoholism or drug abuse within 1 year prior to screening
* History of significant allergies
* Allergy or sensitivity to any of the investigational product ingredients
* Use of medicinal marijuana
* Clinically significant abnormal laboratory results at screening
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  Assessment of blood pressure
Safety Blood Parameters | 8 weeks
  Assessment of safety blood parameters: CBC, electrolytes (Na, K, Cl), kidney function (creatinine), liver function (AST, ALT, GGT and bilirubin)
Heart Rate | 8 weeks
  Assessment of heart rate

SECONDARY OUTCOMES:
Physiological Performance | 8 weeks
  6 Minute Walk Test
Physiological Performance | 8 weeks
  30 Second Chair Stand Test
Physiological Performance | 8 weeks
  Physical Activity Scale for the Elderly
Body Weight | 8 weeks
Blood Pressure | 8 weeks
Serum Glucose | 8 weeks
Lipid Profile | 8 weeks
Quality of Life and Sleep Quality | 8 weeks
  Health Assessment Questionnaire
Quality of Life and Sleep Quality | 8 weeks
  Older People's Quality of Life Questionnaires
Blood NAD+ | 8 weeks

OTHER OUTCOMES:
Expression Profile of Peripheral Blood Mononuclear Cells | 8 weeks
Pain Assessment | 8 weeks
  VAS Pain Scale
Endothelial Function | 8 weeks
  EndoPat

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada